CLINICAL TRIAL: NCT04418115
Title: Acupuncture for Fatigue in Breast Cancer Survivors: a Study Protocol for a Pragmatic, Mixed-method, Randomised Controlled Trial
Brief Title: Fatigue As a Late Effect in Breast Cancer Survivors - is Acupuncture a Treatment Option?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristiania University College (Other)
Collaborators: Norwegian Cancer Society (Other); University of Bergen (Other); Memorial Sloan Kettering Cancer Center (Other); Dana-Farber Cancer Institute (Other); University Hospital, Akershus (Other); University of York (Other); University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AcuBreast 2020
Record Dates: First submitted 2019-11-09; First posted 2020-06-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-06

CONDITIONS: Fatigue; Depression, Anxiety; Insomnia; Hot Flashes; Quality of Life
MeSH Terms: conditions — Fatigue; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Hot Flashes | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The study is a pragmatic, mixed-method, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The statistician is not involved in any other aspect of the study, hence we can secure that the evaluation of the outcomes are done blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture + usual care (Experimental): Participants randomized to acupuncture treatment will receive 12 acupuncture treatments during 8-12 weeks.
  Interventions: Other: Acupuncture; based on Tradidtional Chinese Medicine
- Usual care (No Intervention): Our control group will receive "business as usual". Hence, they will continue with their usual care for their CRF. By inclusion in the study and by the end of it, the participants in the control group will fill in the requested and similar instruments as the participants in the acupuncture group. Further, we will document any medical care they have received during the study period. This includes also life styles advice, and to which point they have followed such advices.

INTERVENTIONS:
Other: Acupuncture; based on Tradidtional Chinese Medicine — Acupuncture is a form of treatment that involves inserting very thin needles through a person's skin at specific points on the body, to various depths. Research suggests that it can help relieve pain, and it is used for a wide range of other complaints.
  Arms: Acupuncture + usual care

SUMMARY:
The success of treatment of breast cancer has improved, hence the prevalence of survivors have increased. However, experienced late effects from the cancer itself or from cancer treatment is substantial. Anti-cancer treatment can have a number of side effects including nausea, fatigue, vomiting, anorexia and alopecia. Late effects such as cancer related fatigue (CRF) are very persistent. CRF is a common side effect of cancer therapy, and affects the quality of life of patients and their families. It is important to point out that CRF is a form of fatigue that are different from normal fatigue which everyone can experience every now and then. Acupuncture is increasingly used in cancer centers both in the US and Europe, and that patients are positive to using acupuncture. Albeit the emerging evidence for acupuncture and CRF, acupuncture has neither been offered as a treatment for CRF within a Norwegian hospital nor in general practice. Hence the investigators think there is a need for a large randomized controlled trial (RCT) in a Norwegian health care setting.

DETAILED DESCRIPTION:
Introduction Breast cancer is the most common tumour type in women worldwide. The success of the treatment of breast cancer have improved hence the prevalence of survivors have increased (American Cancer Society). However, experienced side effects from the cancer itself or from cancer treatments is substantial. Anti-cancer treatment can have a number of side-effects including nausea, fatigue, vomiting, anorexia and alopecia (1 - 3). However, some side effects such as cancer-related fatigue (CRF) are very persistent. CRF is a common adverse effect of cancer and cancer therapy, and effects the quality of life of the patients (4). The definition of CRF from the National Comprehensive Cancer Network (NCCN) is that it is "a distressing, persistent, subjective sense of physical, emotional and/or cognitive tiredness, related to cancer or cancer treatment, that is not proportional to recent activity and interferes with usual functioning" (5). It is important to point out that CRF is a form of fatigue that are different from normal fatigue which everyone can experience every now and then. The symptoms of CRF is under-reported by patients and underestimated and undertreated by clinicians, despite the prevalence and negative impact of CRF (6). It is recommended to patients that they are screened for CRF after completion of primary treatment and that they are offered specific information and strategies for management of the fatigue (7). Getting CRF as a side-effect after cancer treatment can have a major impact in their life.

In Norway on average 3090 women are diagnosed with breast cancer each year, giving a incidence rate per 100 000 persons of 121,0. In 2014, 3348 patients were diagnosed with breast cancer. The prevalence of fatigue is high in breast cancer survivors (BCS), with some studies reporting as many as 50% of the patients experiencing this (8). In a meta-analysis involving 12327 BCS, concluded that approximately one in four BCS suffers from severe fatigue (9). Several different treatments have been recommended for CRF such as exercise, psychosocial intervention, pharmacological interventions and mind-body interventions (4). From several randomized trials mind-body interventions such as yoga and acupuncture has been shown to relieve fatigue in cancer survivors (7). These studies, have however not focused solely on BCS but included other cancer types as well (10). Acupuncture has been shown to have an effect on CRF (10,11). A recent meta-analysis on CRF and acupuncture is positive (12) In Norway BCS are offered treatment such as cognitive behaviour therapy, exercise, relaxation techniques, yoga and nutritional coaching for their CRF. The use of acupuncture in the treatment of chemotherapeutic induced nausea is well established in Norway (13), also a Norwegian study on acupuncture on hot flashes in breast cancer patients has been published (14). The patients are found to be positive to acupuncture (15,16). In US acupuncture seems to have found its place in several hospitals which offers integrative medicine care to cancer patients (10).

Methodological approach A pragmatic, randomised controlled trial At the moment the study group, behind this present application, is running a pilot study on fatigue in breast cancer survivors with acupuncture as the intervention. This pilot study has been approved by the Regional Committee for Medical and Health Research Ethics (REK sør-øst A; reference 2017/2197). The purpose of conducting this pilot study is to examine the feasibility of our approach that is intended to be used in the planned larger randomised controlled study. Hence the design and methodological approach of the study in question wil be equal to the ongoing pilot study. By doing this the investigators can evaluate the feasibility of recruitment, randomization, collaboration, assessment procedures, and implementation of acupuncture. This will help us also to identify, revisions, if any, needed in the design of the larger, pragmatic randomised trial.

The intention with the pragmatic, RCT is to test acupuncture as a complete treatment package, i.e. including the therapeutic relationship and expectation, and address the important question of the overall effect of acupuncture-care, which is highly relevant to breast cancer survivors experiencing CRF. This question concerning the overall effect of acupuncture is also of importance for their health care providers and health authorities in general. As such a pragmatic trial will help users choose between options for care, and ''explanatory'' to describe trials that test causal research hypotheses (i.e., that a given intervention causes a particular benefit).Further, a pragmatic trials are primarily designed to determine the effects of an intervention under the usual conditions in which it will be applied, whereas explanatory trials are primarily designed to determine the effects of an intervention under ideal circumstances.

Baseline assessment includes sociodemographic data, medical and gynaecological history, previous experience with acupuncture, which other self-provided and therapist-provided interventions they have used earlier to relieve fatigue, current use of drugs and dietary supplements, level of physical activity, smoking status and level of alcohol consumption.

At each treatment session the acupuncturists ask specifically about, and record, any adverse events that have occurred during or after the last treatment, and adverse event forms are filled in at 4, 8 and 12 weeks.

Fatigue, and the severity of it, will be measured at inclusion/baseline, just after acupuncture treatment. This will be measured after 12 weeks after the inclusion in the control group; thereafter in both groups at 6 months after baseline evaluation. All secondary measurements will be measured at the same time intervals.

Participants and recruitment Women between 18-60 yrs who are defined as breast cancer survivors by their respective cancer hospital will be invited to take part in the study.To achieve a homogenues group of participants an important inclusion criteria be that they are treated with Tamoxifen. The potential participants will be given written information about the study - no further information will be given by the health personnell at the hospital. If they want to participate, after reading the information, the participants have to sign the paper and send it to Kristiania University College/AcuBreast study by a pre addressed and stamped envelope. Thereafter the research team will contact the potential participants. Women who are interested in participating, will than register their fatigue on a Visual Analog Pain Scale (VAS); women scoring ≥4 will be eligible. Participants will be excluded if they have needle phobia; low platelet count (<50 000); co-morbidity with a bleeding disorder; co-morbidity with thyroid dysfunction; planned to be pregnant during the study period or present pregnant; haemoglobin levels <10 g/dl and haematocrit <30; anaemia on active pharmacological treatment or receiving blood transfusion or steroids, and life expectancy <6 months. In addition, lymphoedematous limbs are excluded from needling.

Randomization Our collaborating statistician from the University of Bergen, will prepare the randomisation database and acts as a central randomisation service.

Acupuncture group The women randomized to acupuncture treatment will receive 12 acupuncture treatments during 8-12 weeks. The participating acupuncturists must have finished their Bachelor degree in acupuncture at least 5 years ago and they will be members of the "The Norwegian Acupuncture Association". The form of acupuncture used in this trial will be based upon theories from Traditional Chinese Medicine (TCM). The diagnostic process in TCM is complex and unique. It is a procedure that guides the practitioners to establish for themselves a correct treatment according to their theoretical knowledge and clinical experience within Chinese medicine. Taking a medical history according to TCM theories, match somehow the experience of a ''lived body.'' Hence added to the acupuncture treatment, there could be given relevant advices in relation to diet, exercise, rest and sex. Such advices are common within TCM; all advices given would be registered within the study in question.

Control group Our control group will do "business as usual". Hence they will continue with their usual care for their CRF. By inclusion in the pilot study and by the end of it, the participants in the control group will fill in the requested and similar instruments as the participants in the acupuncture group.

Safety of acupuncture and special procedures for our patient group. Acupuncture in general has been reported to be safe in the hands of well-educated acupuncturists (17-19). Special precautions have been described for treating cancer patients with acupuncture (20). Avoid needling the arm of patients who have undergone axillary dissection, the same applies for any lymphedematous limbs. Possible participants with low platelet count; comorbidity with a bleeding disorder or are planning pregnancy within the study period will be excluded.

Data analysis All analyses will be conducted blinded to group allocation. The primary analysis is intention-to-treat, comparing mean changes from baseline to end of treatment after 12 weeks in the two groups, using a two-sample t-test. In the presence of meaningful baseline differences, analysis of covariance will be employed. It is anticipated that the data will be somewhat right-skewed, therefore analyses will be checked after appropriate data conversion, and also checked using non-parametric methods. Secondary analyses will compare the changes at different time points. Secondary measures will be analyzed using appropriate parametric or non-parametric methods. Subgroup analyses include per-protocol analyses to assess efficacy of acupuncture care, and comparison of changes in fatigue scores among women grouped by TCM syndromes.

Data and safety monitoring The study is performed according to the Helsinki declaration and Good Clinical Practice requirements. Application for approval of the studies will be sent to the Regional Committee for Medical and Health Research Ethics (REK sør-øst).

Dissemination and communications strategy The investigators will utilize dissemination and public outreach to boost the impact of the work in the research project. Scientific results will be published in high-impact journals, and results will be presented on national and international scientific meetings.

Project management Professor Terje Alraek, at Kristiania University College, Institute of Health Sciences, has worked within the field of acupuncture for more than 30 years. First and still as a clinician and from 1994 has he been involved in research on acupuncture. He has during his research initiated, been invited to and developed several international groups of researcher with interest in acupuncture. Alraek and the foreign members of the established research group have published a substantial amount of scientific papers and they have also published many books in relation to all the problems of doing research on such a complex intervention as acupuncture.

The research team are happy to have managed to have one national- and two important international cancer centers as collaborating partners on this project. Our collaborating partners in US besides being researchers, are also experienced clinicians in treating breastcancer survivors with acupuncture for fatigue at their respective centers.

User involvement The user representative has a special responsibility for ensuring that the research is in line with the preferences, values and needs of breast cancer patients suffering from CRF.

Qualitative studies Participants from, the acupuncture- and control groups, will be asked to write about their experiences. The former with acupuncture treatment and the latter one of being in the control group.

Biomarkers and Cancer related fatigue Nested within this RCT, is one sub-study measuring biomarkers (CRP, IL1, IL6, TNF-α, CRP, aPL in addition to the current genotype genes TNF-308 and IL-6-174) from blood samples (n=80). Such biomarkers can potentially address changes of cancer related fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer survivors, aged 18 or older, not receiving any curative cancer treatment
2. Fatigue score on a VAS scale ≥4 will be eligible
3. Sufficient knowledge of Norwegian is necessary for communicating with the acupuncturist and for filling in and understanding all the Norwegian questionnaires within the study.
4. Participants who have freely agreed to take part in the study and have signed an informed consent form.

Exclusion Criteria:

1. Any causal pathology related to fatigue or receiving ongoing acupuncture treatment for fatigue.
2. Participants who are pregnant at baseline or planning to get pregnant within the treatment period will be excluded. Reason is that several acupuncture points should be avoided during pregnancy and several of those are related to the treatment of fatigue.
3. Potential participants who are unable to understand, speak, or who find it difficult to communicate in Norwegian will be excluded from the study.
4. Individuals presenting with clinically diagnosed conditions or pathologies known to contribute to fatigue and persons whose fatigue could be attributed to pre-existing conditions

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Fatigue | 12 weeks (treatment completion), Change from baseline registration at 3 and 6 month
  Chalders Fatigue questionnaire (FQ)
Fatigue 2 | Change from baseline registration at 3 and 6 month
  Fatigue Severity Scale (FSS)

SECONDARY OUTCOMES:
Anxiety and depression | 12 weeks (treatment completion), Change from baseline registration at 3 and 6 months
  Hospital and Anxiety Depression scale (HADS). The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. Scores are constructed by summation, whereby increasing scores indicate increasing burden. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Bergen Insomnia Scale | 12 weeks (treatment completion), Change from baseline registration
  The Bergen Insomnia Scale consist of six items, of which the first three pertain to sleep onset, maintenance, and early morning wakening insomnia, respectively. The last three items refer to not feeling adequately rested, experiencing daytime impairment, and being dissatisfied with current sleep. Each item is rated on an 8-point scale, ranging from 0 to 7 days per week. A total composite score is calculated by adding together the scores for each item, yielding a total score with a possible range of 0 to 42. A high score indicating more severe problems.
The Epworth Sleepiness Scale | 12 weeks (treatment completion), Change from baseline registration
  The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3). The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Hot flashes | 12 weeks (treatment completion), Change from baseline registration
  Self-managed diary reporting the frequency and the severity of hot flashes
Quality of Life (QLQ) questionnaire | 12 weeks (treatment completion), Change from baseline registration
  EORTC QLQ-C30,
Quality-adjusted life year - QALY questionnaire | Baseline and 6 months
  EQ-5D- 5L

CONTACTS AND LOCATIONS:
Overall Officials: Terje Alraek, PhD, Principal Investigator — School of Health Sciences, Kristiania University College
Locations (1):
- Kristiania University College, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Baseline data, primary and secondary outcomes may be shared. This is applicable since all data sheets are rendered anonymous by removing participant names and addresses. Trial number alone identifies all computerized data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2024 and for 3 years
Access Criteria: Application to the sent to the Principle Investigator

REFERENCES:
- [Derived] Alraek T, Skjerve H, Sorensen A, Lie SA, Presterud Odegard H, Lu W, Mao J, Deng G, Lee MS, Birch S, Lamu AN, Kim TH, MacPherson H. Acupuncture for fatigue in breast cancer survivors: a study protocol for a pragmatic, mixed method, randomised controlled trial. BMJ Open. 2024 Jul 30;14(7):e077514. doi: 10.1136/bmjopen-2023-077514. PMID 39079925